CLINICAL TRIAL: NCT02290704
Title: Changes of Retinal Oxygen Saturation in Patients With Graves' Ophthalmopathy Under Different Managing Conditions and in Normal People
Brief Title: Retinal Oxygen Saturation in Patients With Graves' Ophthalmopathy and in Normal People
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiaonan Yang, the graduate student of Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: 2013MEKY039
Record Dates: First submitted 2014-11-03; First posted 2014-11-14 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Graves' Ophthalmopathy
Keywords: oxygen saturation; retinal vessels; thyroid associated ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- controls: People without eye disease
- GO patients: patients with Graves' ophthalmopathy

SUMMARY:
Find if the retinal function is affected in both the nonsevere and the severe stage of Graves' ophthalmopathy (GO) by comparing the retinal oxygen saturation of GO patients with that of normal people.

DETAILED DESCRIPTION:
Graves'ophthalmopathy (GO), also called thyroid-associated ophthalmopathy, is often mild and self-limiting, and probably declining in frequency, with only 3-5% of cases posing a threat to eyesight, remaining a pathogenetic enigma and a therapeutic dilemma. In its nonsevere expression, the symptoms and signs include Photophobia, Foreign body sensation, Eyelid retraction, increased intraocular pressure, Lagophthalmos, and Mild diplopia. In its severe expression, it is a disfiguring and invalidating disease with the optic nerve damaged. However, in this study, we want to find if the retinal vessels is affected in the early stage of the disease through observing the oxygen saturation of the retinal vessels and compare it with that of the normal people.

ELIGIBILITY:
Inclusion Criteria for GO patients:

1. conforms to the diagnosis of Graves' ophthalmopathy;
2. age > 18;
3. volunteered to participate in this research, and sign the informed consent.

Inclusion Criteria for Control group:

1. age > 18;
2. diopter within + / - 3D;
3. volunteered to participate in this research, and sign the informed consent.

Exclusion Criteria for GO patients:

1. Fundus could not be seen clearly;
2. pregnant and lactating women;
3. could not tolerate the examination.

Exclusion Criteria for Control group:

1. with severe systemic disease and cause eye lesions;
2. have history of eye disease, ocular trauma and eye surgery impacting on visual function;
3. pregnant and lactating women;
4. could not tolerate the examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Controls- normal people; GO patients- patients with Graves' ophthalmopathy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
changes of retinal oxygen saturation in patients with GO under different managing conditions | before surgery ( or glucocorticoids administration), 1 week and 4 weeks after surgery ( or glucocorticoids administration)

CONTACTS AND LOCATIONS:
Overall Officials: Danping Huang, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University; Xiaonan Yang, Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University; Siming Ai, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University; Huasheng Yang, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Bahn RS, Heufelder AE. Pathogenesis of Graves' ophthalmopathy. N Engl J Med. 1993 Nov 11;329(20):1468-75. doi: 10.1056/NEJM199311113292007. No abstract available. PMID 8413459
- [Background] Alford EL, Soparkar CN. Management of the 'tight orbit' and associated visual loss. Curr Opin Otolaryngol Head Neck Surg. 2013 Aug;21(4):417-22. doi: 10.1097/MOO.0b013e32836312a1. PMID 23838551
- [Result] Michelson G, Scibor M. Intravascular oxygen saturation in retinal vessels in normal subjects and open-angle glaucoma subjects. Acta Ophthalmol Scand. 2006 Jun;84(3):289-95. doi: 10.1111/j.1600-0420.2005.00631.x. PMID 16704685